CLINICAL TRIAL: NCT07017179
Title: A Phase IIa Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of AZD6234, AZD9550, and AZD6234 in Combination With AZD9550 in Chinese Participants Living With Obesity/Overweight
Brief Title: This is a Multi-centre, Multi-drug, Platform Study in Chinese Participants Living With Obesity / Overweight
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D8750C00009
Record Dates: First submitted 2025-05-14; First posted 2025-06-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Obesity/Overweight
Keywords: Obesity; Overweight; Chinese Participants; AZD6234; AZD9550
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- AZD6234 (sub-study 1) (Experimental): Participants will receive subcutaneous injection of AZD6234 on Day 1 and continue for 16 weeks.
  Interventions: Drug: AZD6234
- Placebo (sub-study 1) (Placebo Comparator): Participants will receive subcutaneous injection of matched volume of placebo on Day 1 and continue for 16 weeks.
  Interventions: Drug: Placebo
- AZD9550（sub-study 2 Cohort A) (Experimental): Participants will receive subcutaneous injection of AZD9550 on Day 1 and continue for 28 weeks.
  Interventions: Drug: AZD9550
- Placebo (sub-study 2 Cohort A) (Placebo Comparator): Participants will receive subcutaneous injection of matched volume of placebo on Day 1 and continue for 28 weeks.
  Interventions: Drug: Plocebo
- AZD6234 in combination with AZD9550 (sub-study 2 Cohort B) (Experimental): Participants will receive subcutaneous injection of AZD6234 and AZD9550 on Day 1 and continue for 28 weeks.
  Interventions: Drug: AZD6234 in combination with AZD9550
- Placebo (sub-study 2 Cohort B) (Placebo Comparator): Participants will receive subcutaneous injection of matched volume of placebo on Day 1 and continue for 28 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD6234 — Participants will receive a subcutaneous injection weekly
  Arms: AZD6234 (sub-study 1)
Drug: Placebo — Participants will receive a subcutaneous injection weekly.
  Arms: Placebo (sub-study 1)
Drug: AZD9550 — Participants will receive a subcutaneous injection weekly
  Arms: AZD9550（sub-study 2 Cohort A)
Drug: Plocebo — Participants will receive a subcutaneous injection weekly
  Arms: Placebo (sub-study 2 Cohort A)
Drug: AZD6234 in combination with AZD9550 — Participants will receive a subcutaneous injection weekly
  Arms: AZD6234 in combination with AZD9550 (sub-study 2 Cohort B)
Drug: Placebo — Participants will receive a subcutaneous injection weekly
  Arms: Placebo (sub-study 2 Cohort B)

SUMMARY:
This study is to assess the safety and tolerability, PK characterisation, efficacy, and immunogenicity of the study intervention, and it allows assessment of the monotherapy or combination therapy of AZD6234 and AZD9550 in different sub-studies.

DETAILED DESCRIPTION:
This is a Phase Ⅱa, multi-centre, multi-drug, platform study in Chinese participants living with obesity/overweight. This platform study will consist of several sub-studies. Eligible participants will be allocated to one sub-study to receive the study intervention(s). Each sub-study will consist of a screening period, a treatment period, and a follow-up period.

Sub-study 1: AZD6234 Monotherapy This study will explore the safety, tolerability, pharmacokinetic (PK), efficacy, and immunogenicity of AZD6234 in Chinese participants with obesity/overweight, approximate 18 participants will be randomised in sub-study 1. The sub-study will comprise 3 periods totalling up to approximately 23 weeks.

Sub-study 2: AZD9550 Monotherapy and AZD6234 in combination with AZD9550 This study will explore the safety, tolerability, PK, efficacy, and immunogenicity of AZD9550 and of AZD6234 in combination with AZD9550 in Chinese participants with obesity/overweight, approximately 30 participants will be randomised in sub-study 2 (15 in Cohort A and 15 in Cohort B). The sub-study will comprise 3 periods totalling up to approximately 35 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 55 years.
2. BMI ≥ 27 kg/m2.
3. Stable body weight for 3 months prior to screening.
4. Male and female (Contraceptive use by participants or participant partners should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies).
5. Participants should refrain from blodd donation throughout the sub-study, including the follow-up period.
6. Negative pregnancy test at screening and randomisation for FOCBP and must not be breastfeeding.

Exclusion Criteria:

1. Have received prescription medication or non-prescription medication for weight loss within the last 3 months prior to screening.
2. History of type 1 or type 2 diabetes mellitus or symptoms indicative of insulinopenia or poor glucose control.
3. Treatment with diabetes medication in past 3 months prior to screening.
4. HbA1c ≥ 6.5% (48 mmol/mol) at screening.
5. Gastroparesis (or similar) requiring treatment.
6. Significant inflammatory bowel disease or other severe disease or surgery affecting the upper GI tract.
7. Significant hepatic disease (except for non-alcoholic steatohepatitis or non-alcoholic fatty liver disease without portal hypertension or cirrhosis) and/or participants with any of the following results at screening:

   1. AST ≥ 2.5 × ULN
   2. ALT ≥ 2.5 × ULN
   3. TBL ≥ 1.5 × ULN.
8. Prior history of cholecystectomy or untreated cholelithiasis.
9. History of acute or chronic pancreatitis or pancreatic amylase or lipase > 2 × ULN at screening.
10. Severely uncontrolled hypertension defined as systolic BP ≥ 160 mmHg and/or diastolic BP ≥ 100 mmHg on the average of 2 seated measurements after being at rest for at least 5 minutes.
11. HR < 50 bpm or > 100 bpm after being at rest for 5 minutes.
12. Impaired renal function defined as eGFR ≤ 45 mL/minute/1.73 m2 at screening (GFR estimated according to CKD-EPI).
13. History of psychosis or bipolar disorder.
14. Severe vitamin D deficiency defined as a 25-OH vitamin D level < 12 ng/mL.
15. Uncontrolled thyroid disease, defined as TSH > ULN or < LLN for the laboratory reference range, as judged by the PI at screening.

    Sub-study 2 only
16. Personal or family history (first-degree relative) of MTC or MEN2.
17. History of marijuana or THC use within 3 months before screening, or unwilling/unable to abstain from marijuana or THC use during the study.
18. Previous hospitalisation for any psychiatric reason.
19. PHQ-9 score ≥ 15 within the 2 years prior to screening or at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 871 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-08-06 (Estimated); Study Completion 2026-08-06 (Estimated)

PRIMARY OUTCOMES:
Numbers of participant with Adverse Events (AEs) and Serious adverse events (SAEs) (sub-study 1). | From baseline to Day 141
  To assess the safety and tolerability of repeated subcutaneous(SC) doses of AZD6234 compared to placebo.
Numbers of participant with Adverse Events (AEs) and Serious adverse events (SAEs) (sub-study 2). | From baseline to Day 225
  To assess the safety and tolerability of repeated SC doses of AZD9550 and AZD6234 in combination with AZD9550 compared to placebo.

SECONDARY OUTCOMES:
PK parameters : Cmax (sub-study 1) | Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 85,106,113,120,127,141 Pre-dose. Day 1,36,43,57,106 post-dose 2,4,8,12,24,36,48,60,72,96 hours.
  To characterise the PK of AZD6234 following repeated subcutaneous (SC) doses.
PK parameters : Tmax (sub-study 1) | Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 85,106,113,120,127,141 Pre-dose. Day 1,36,43,57,106 post-dose 2,4,8,12,24,36,48,60,72,96 hours.
  To characterise the PK of AZD6234 following repeated SC doses.
PK parameters : AUClast (sub-study 1) | Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 85,106,113,120,127,141 Pre-dose. Day 1,36,43,57,106 post-dose 2,4,8,12,24,36,48,60,72,96 hours.
  To characterise the PK of AZD6234 following repeated SC doses.
PK parameters : AUCtau (sub-study 1) | Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 85,106,113,120,127,141 Pre-dose. Day 1,36,43,57,106 post-dose 2,4,8,12,24,36,48,60,72,96 hours.
  To characterise the PK of AZD6234 following repeated SC doses.
Percent change in body weight from baseline to Week 16 (sub-study 1) | From baseline to Week 16
  To assess the effects of AZD6234 on the body weight change from baseline with and without placebo correction.
Incidence of ADA to AZD6234 (sub-study 1). | Day 1 to Day 141
  To evaluate the immunogenicity of AZD6234 following repeated SC doses.
ADA titer of AZD6234 (sub-study 1). | Day 1 to Day 141
  To evaluate the immunogenicity of AZD6234 following repeated SC doses.
PK parameters : Cmax (sub-study 2 Cohort A) | Days 1, 15, 29, 57, 85, 113, 141, 190, 204, 211, 225 per dose. Days 1, 57, 113, 141,190 post-dose 6, 12, 18, 24 hours (± 10 minutes). Day 190 post-dos 30, 36, 42, 48, 54, 60, 72, 96, 120, 144,168 hours (± 30 minutes).
  To characterise the PK of AZD9550 following repeated SC doses.
PK parameters : Tmax (sub-study 2 Cohort A) | Days 1, 15, 29, 57, 85, 113, 141, 190, 204, 211, 225 per dose. Days 1, 57, 113, 141,190 post-dose 6, 12, 18, 24 hours (± 10 minutes). Day 190 post-dos 30, 36, 42, 48, 54, 60, 72, 96, 120, 144,168 hours (± 30 minutes).
  To characterise the PK of AZD9550 following repeated SC doses.
PK parameters : AUClast (sub-study 2 Cohort A) | Days 1, 15, 29, 57, 85, 113, 141, 190, 204, 211, 225 per dose. Days 1, 57, 113, 141,190 post-dose 6, 12, 18, 24 hours (± 10 minutes). Day 190 post-dos 30, 36, 42, 48, 54, 60, 72, 96, 120, 144,168 hours (± 30 minutes).
  To characterise the PK of AZD9550 following repeated SC doses.
PK parameters : AUCtau (sub-study 2 Cohort A) | Days 1, 15, 29, 57, 85, 113, 141, 190, 204, 211, 225 per dose. Days 1, 57, 113, 141,190 post-dose 6, 12, 18, 24 hours (± 10 minutes). Day 190 post-dos 30, 36, 42, 48, 54, 60, 72, 96, 120, 144,168 hours (± 30 minutes).
  To characterise the PK of AZD9550 following repeated SC doses.
Plasma trough concentration (sub-study 2 Cohort B). | Day 1 to Day 225
  To characterise the PK of AZD9550 and AZD6234 following repeated SC doses
Percent change in body weight from baseline to Week 28 (sub-study 2 ), placebo as comparator | From baseline to Week 28
  To assess the effects of AZD9550 and AZD6234 in combination with AZD9550 on the body weight change from baseline with and without placebo correction.
Percent change in body weight from baseline to Week 28 (sub-study 2, AZD9550 as comparator) | From baseline to Week 28
  To assess the effects of AZD6234 in combination with AZD9550 compared to AZD9550 on the body weight change from baseline.
Incidence of ADA to AZD9550 (sub-study 2). | Day 1 to Day 225
  To evaluate the immunogenicity of AZD9550 following repeated SC doses.
ADA titer of AZD9550 (sub-study 2 Cohort A). | Day 1 to Day 225
  To evaluate the immunogenicity of AZD9550 following repeated SC doses.
Incidence of ADA to AZD6234 and AZD9550 combination therapy (sub-study 2 Cohort B). | Day 1 to Day 225
  To evaluate the immunogenicity of AZD6234 and AZD9550 following repeated SC combination therapy doses.
ADA titer of AZD6234 and AZD9550 combination therapy (sub-study 2 Cohort B). | Day 1 to Day 225
  To evaluate the immunogenicity of AZD6234 and AZD9550 following repeated SC combination therapy doses.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Research Site, Jinan
  - Research Site, Nanjing
  - Research Site, Shanghai